CLINICAL TRIAL: NCT00234208
Title: A Randomized Controlled Study of Early Mini-invasive Medical Thoracoscopy Versus Simple Chest Tube Drainage in Complicated Parapneumonic Effusions or Pleural Empyema - ESMITE (European Study on Mini-invasive Thoracoscopy in Empyema)
Brief Title: Early Medical Thoracoscopy Versus Simple Chest Tube Drainage in Complicated Parapneumonic Effusion and Pleural Empyema
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Lancardis Foundation (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK 186/05
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Complicated Parapneumonic Effusion; Pleural Empyema
Keywords: Complicated parapneumonic effusion; Pleural empyema; Intervention; Medical thoracoscopy; Chest tube drainage
MeSH Terms: conditions — Empyema, Pleural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical thoracoscopy (Experimental)
  Interventions: Procedure: Medical thoracoscopy
- Simple chest tube drainage (Active Comparator)
  Interventions: Procedure: Simple chest tube drainage

INTERVENTIONS:
Procedure: Medical thoracoscopy
  Arms: Medical thoracoscopy
Procedure: Simple chest tube drainage
  Arms: Simple chest tube drainage

SUMMARY:
Multicenter, randomized controlled study to compare early mini-invasive thoracoscopy to simple chest tube drainage in complicated parapneumonic effusions or pleural empyema. 100 patients will be recruited. Follow-up will be 3 months. It will be looked at the rate medical cure, the need for secondary interventions, death and duration of hospital stay. In a nested trial in 20 patients the intrapleural pharmacokinetics of linezolid (approved antibiotic agent) will be measured.

DETAILED DESCRIPTION:
Background Pleural empyema has a high morbidity and mortality. Until now it is not clear which method is best to initially drain the pus, especially in complicated effusions with septa.

The objective of this study is to compare the standard treatment of simple chest tube drainage to early mini-invasive medical thoracoscopy. In earlier studies medical thoracoscopy has been a safe and effective method in pleural diseases. However there is no prospective data available.

Methods We conduct a prospective randomized controlled multicenter study on 100 patients with complicated parapneumonic effusions with septa or empyema with frank pus. Patients will be randomized to receive either simple chest tube drainage or early medical thoracoscopy. The latter will be performed in local anaesthesia and analgosedation according to the standards set by the European Study on Medical Video-Assisted Thoracoscopy (ESMEVAT)-group. Fibrinolysis will be used routinely. In 20 patients a nested study on the intrapleural pharmacokinetics of linezolid as antibiotic agent will be performed.

Follow-up will be structured on day 1, day 7, before discharge and after 3 months including chest radiographs and clinical and laboratory evaluations.

Outcome Primary outcome will be medical cure without the need of secondary intervention or death.

As secondary outcome we will measure duration of hospital stay, adverse events.

Provisional agenda Start of study: October 2005 End of study: October 2007

Potential outcome & benefit The study should clarify the role of early medical thoracoscopy in patients with complicated parapneumonic effusions or pleural empyema. Different authors have speculated that early intervention could be preferable. On the other hand, in many centres worldwide patients are primarily treated by a simple chest tube with or without pleural fibrinolysis. In case of failure of simple drainage, but this means several "precious" days later, a more invasive procedure is needed. At that moment tight pleural septa have formed, and often a surgical VATS or thoracotomy in general anaesthesia becomes necessary. Therefore, this pivotal study could lead to changes in the management of patients with pleural empyema.

ELIGIBILITY:
Inclusion Criteria:

* Septated pleural effusion (ultrasonography) in the context of a lower respiratory tract infection
* Frank pleural empyema (pus)

Exclusion Criteria:

* Fibrothorax
* Tuberculous empyema
* Medical thoracoscopy cannot be performed within 24 hours
* Pregnancy
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Medical cure without secondary Intervention
Death

SECONDARY OUTCOMES:
Duration of hospital stay
Radiological outcome
Duration of drainage
Total amount of drainage fluid
Estimated cost
Adverse events
Pleural pharmacokinetics of linezolid

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Brutsche, MD, Prof., Principal Investigator — Pneumology, Kantonsspital St. Gallen
Locations (5):
- Department of Pneumology, University Hospital of Alexandroupolis, Alexandroupoli, Greece
- Italy (3):
  - Pulmonology Unit, Spedali Civili di Brescia, Brescia
  - UO Pneumologia, Imperia
  - Pulmonology and Thoracic Endoscopy Unit Azienda Ospedaliera di Parma, Parma
- Centre Valaisan de Pneumologie, Crans-Montana, Switzerland